CLINICAL TRIAL: NCT06717165
Title: A Randomized, Double-Blind, Clinical Trial to Study the Efficacy and Mechanisms of Transcranial Alternating Current Stimulation (tACS) Concurrent With Exposure-based Cognitive-Behavioral Therapy (CBT) for Obsessive-Compulsive Disorder (OCD)
Brief Title: Efficacy and Mechanism of Augmentation of Cognitive Behavioral Therapy With Transcranial Alternating Current Stimulation(tACS) for Obsessive-Compulsive Disorder (OCD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Zhen Wang, vice-president, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMHC-OCD-013
Record Dates: First submitted 2024-12-01; First posted 2024-12-04 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Obsessive Compulsive Disorder (OCD)
Keywords: cognitive-behavioral therapy; exposure and response prevention; transcranial alternating current stimulation
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tACS+exposure based CBT (Active Comparator): The exposure and response prevention (ERP) treatment concurrently with an anode transcranial alternating current stimulation over the mPFC will be applied 8 times (tACS+ERP, 8 sessions) in the whole treatment.
  Interventions: Combination Product: ERP combined with high-definition active tACS
- sham tACS +exposure based CBT (Sham Comparator): the exposure and response prevention (ERP) treatment concurrently with an sham transcranial alternating current stimulation over the mPFC will be applied 8 times (sham tACS+ERP, 8 sessions) in the whole treatment.
  Interventions: Combination Product: ERP combined with sham tACS

INTERVENTIONS:
Combination Product: ERP combined with high-definition active tACS — The active tACS +ERP referred to a period of tACS applied in the first 20 minutes of the ERP treatment (the tACS device was activated when ERP began and deactivated automatically while ERP continued). The total treatment phase lasted eight weeks and included ten sessions with experienced psychotherapists following a specific manual for the tACS+ERP treatment. Based on the EEG parameters, individualized modeling was conducted to determine specific stimulation parameter schemes (stimulation frequency). Anode electrode will be localized in front of the mPFC on the Fz point according to the EEG international reference. Four cathode electrodes will be placed around (i.e. AFz, Fcz, F1, F2).
  Arms: active tACS+exposure based CBT
Combination Product: ERP combined with sham tACS — Patients will get the same CBT setting as the active tACS group and they were applied the sham tACS cocurrently with ERP. The sham tACS device is the same as the active comparator's except that the sham tACS will only deliver a current stimulation for the first and last 15 seconds in order to produce somatic sensation in patients similar to that induced by the active tACS.
  Arms: sham tACS +exposure based CBT

SUMMARY:
This study aims to evaluate the feasibility and clinical outcome of the Exposure-based Cognitive-Behavioral Therapy (CBT) concurrent with Transcranial Alternating Current Stimulation (tACS) using individualized stimulation frequency in treating obsessive-compulsive disorder (OCD) patients, and explores the potential neural mechanisms of treatment effect by magnetic resonance imaging (MRI) and electroencephalography (EEG).

DETAILED DESCRIPTION:
The current study aims to evaluate feasibility and clinical outcome of exposure-based CBT (ERP) combined with tACS over the prefrontal cortex (mPFC) in treatment of OCD patients. 62 OCD patients will be randomized into two groups (ERP+active tACS, ERP+sham tACS stimulation). All patients will be received 10 sessions of individual ERP in a two-month period, including 8 sessions of concurrent tACS with ERP (tACS+ERP). Based on the EEG parameters, individualized modeling was conducted to determine specific stimulation parameter schemes (stimulation frequency).

The treatment program consists of a total of 10 sessions, with the first and last sessions being psychological therapy only. The middle eight sessions will involve concurrent transcranial alternating current stimulation (tACS) and exposure and response prevention (ERP). The timing of assessments is designed to capture changes in symptom severity during the intervals between consecutive combined treatment sessions.

Three independent evaluators will assess the severity of patients' obsessive-compulsive symptoms using the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) at four time points:

Baseline assessment (prior to the start of treatment); After the first combined session (Session 2) and before the second combined session (Session 3); After the fourth combined session (Session 5) and before the fifth combined session(Session 6); After the eighth combined session (Session 9) and before the final treatment session (Session 10).

Patients will also undergo electroencephalography (EEG) assessments at each evaluation time point. The current study aims to explore whether the administration of individualized stimulation frequency tACS in conjunction with ERP can enhance the efficacy of ERP, providing early evidence for revealing the potential neural mechanisms underlying this treatment. Additionally, participants will undergo magnetic resonance imaging (MRI) scans at treatment baseline and after the completion of the full course of treatment.

ELIGIBILITY:
The investigators recruited outpatient adults with OCD confirmed by the Mini-International Neuropsychiatric Interview (MINI). The following inclusion and exclusion criteria were also applied:

Inclusion Criteria:

* 18-60 years old
* With at least 9 years of education
* Y-BOCS score ≥16
* No history of serious medical, neurological illness or other psychotic disorders other than OCD (anxiety or mild to moderate depression secondary to OCD was not exclusionary)
* Medication-free or had received stable medication for at least 8 weeks before entering the study and continued the same medication throughout the study

Exclusion Criteria:

* History of serious medical, neurological illness or other psychotic disorders other than OCD
* OCD symptoms are severe, preventing the patient from completing the required assessment and examination
* Serious suicide risk
* Women who are pregnant or planning to become pregnant
* Currently taking antiepileptic medication
* Clinically significant physical illnesses or laboratory test abnormalities that have clinical significance
* Previous completion of a full course of CBT/ERP treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To explore the differences in treatment efficacy between active and sham transcranial alternating current stimulation (tACS) concurrent with exposure and response prevention (ERP)(tACS+ERP) in patients with obsessive-compulsive disorder (OCD). | baseline, 2weeks, 4weeks,8 weeks (baseline, after Session 2, 5, 10)
  The primary outcome measure of this study is the change in Yale-Brown Obsessive Compulsive Scale (Y-BOCS) scores from baseline at the completion of the 8th tACS + ERP treatment.
  Yale-Brown Obsessive Compulsive Scale (Y-BOCS)：The total score of the scale ranges from 0 to 40, with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, PhD, MD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China